CLINICAL TRIAL: NCT03632525
Title: A Pilot Trial of Intravenous Iron for the Treatment of Iron Deficiency in Adult Patients With Cystic Fibrosis
Brief Title: Intravenous Iron in Adults With Cystic Fibrosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PID12800
Record Dates: First submitted 2018-06-21; First posted 2018-08-15 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Cystic Fibrosis; Iron-deficiency
MeSH Terms: conditions — Cystic Fibrosis; Anemia, Iron-Deficiency | interventions — ferric carboxymaltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intravenous iron (Experimental): All participants will receive a single dose of intravenous ferric carboxymaltose
  Interventions: Drug: Ferric carboxymaltose

INTERVENTIONS:
Drug: Ferric carboxymaltose — Single dose of 20 mg/kg ferric carboxymaltose (maximum 1000 mg for patients with haemoglobin <14 g/dL or 500 mg for patients with haemoglobin ≥14 g/dL).
  Other Names: Ferrinject

SUMMARY:
This pilot interventional cohort study will examine the effects of intravenous iron in adults with cystic fibrosis and iron deficiency.

DETAILED DESCRIPTION:
Iron deficiency is common in adults with cystic fibrosis, and is associated with adverse outcomes. Oral iron supplementation is poorly tolerated and may be ineffective. In some centres, intravenous iron is used to correct iron deficiency, but concerns have been raised about the safety of this treatment in the setting of chronic airways infection. The investigators are therefore planning a pilot interventional cohort study examining the effects of intravenous iron in a group of adults with cystic fibrosis. Patients will be recruited in Oxford and studied prospectively over 16 weeks, with iron given at week 4. The primary focus of this single-centre pilot/feasibility study is safety, specifically in relation to infection.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years with established diagnosis of cystic fibrosis
* Iron deficiency (transferrin saturation ≤16 % or ferritin <15 μg/l, within last 4 months)

Exclusion Criteria:

* Urgent (<6 weeks) need for iron supplementation
* Active infection (currently requiring IV antibiotics)
* Previous intravenous iron supplementation (within last 4 months)
* Current oral iron supplementation
* Hypersensitivity to ferric carboxymaltose
* Active non-tuberculous mycobacterial pulmonary disease (as defined by ATS-IDSA criteria)
* Liver failure
* Ferritin >300 μg/l or transferrin saturation >45%
* Pregnancy or breast feeding
* Previous transplantation
* Judged by member of trial team to be unlikely to comply with safety aspects of trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
Incidence of new infective events during 4 weeks before intravenous iron, compared with 4 weeks after intravenous iron | 8 weeks
  New infective events are defined as any of:
  1. New microbiological isolate on routine sputum culture (organism not cultured in 12 months prior to study)
  2. Clinical infection requiring IV antibiotics (as determined by clinical team)
  3. Admission to hospital for infection-related reason (as determined by clinical team)
  4. Significant deterioration in lung function (>10% fall in FEV1), not otherwise explained (as determined by clinical team)

SECONDARY OUTCOMES:
Incidence of new infective events during 12 weeks before intravenous iron, compared with 12 weeks after intravenous iron | 16 weeks (plus 8 weeks of retrospective data collection from notes)
  Infective events are defined as per primary outcome. Data relating to the 8 weeks prior to the 16-week prospective study period will be obtained from the medical records.
Change in number of antibiotic days | 16 weeks
  Assessed by review of clinical notes and patient self-reporting, to determine total number of days on which the patient was treated with antibiotics
Change in abundance of sputum Pseudomonas | 16 weeks
  Assessed by quantitative PCR
Change in sputum microbiological diversity | 16 weeks
  Assessed by microbiota analysis (16s rRNA gene sequencing)
Change in exercise capacity (shuttle walk test) | 16 weeks
  Standardised and validated exercise test involving exercise at progressive intensity
Change in lung function (FEV1) | 16 weeks
  Assessed by spirometry
Change in arterial oxygen saturation | 16 weeks
  Assessed by non-invasive pulse oximetry
Change in body mass index | 16 weeks
  Calculated by standard formula: BMI=weight/(height squared)
Change in quality of life (CFQ-R questionnaire) | 16 weeks
  The Cystic Fibrosis Questionnaire-Revised (CFQ-R) is a 48-item questionnaire that provides scores in twelve quality of life domains (physical functioning, vitality, emotional state, social limitations, role limitations, embarrassment, body image, eating disturbance, treatment constraints) and three symptom domains (respiratory, digestive, weight). Scores ranging from 0 to 100 are calculated for each quality of life domain, using a published method, where a higher score indicates a more favourable health status.
Change in quality of life (SF-36 questionnaire) | 16 weeks
  The 36-item short form questionnaire (SF-36) provides scores in eight major domains of health (physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions). Each is scored on a scale from 0-100, where a higher value represents a more favourable health status. The domains may be combined to provide two summary scores, namely the 'physical component summary' and the 'mental component summary', each of which is also scored from 0-100. In calculating the respective summary scores, subscales related to physical or psychological health (as appropriate) are positively weighted, according to a published method.
Change in pulmonary artery pressure, assessed by echocardiography (exploratory outcome) | 16 weeks
  Assessed via changes in tricuspid regurgitant jet velocity
Percentage of eligible patients entering and completing the study | 16 weeks
  Calculated based on number of eligible patients that enter and/or complete the study.
Percentage of patient in whom each outcome is successfully measured | 16 weeks
  Calculated based on number of participating patients in whom each outcome is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Nick P Talbot, BMBCh DPhil, Principal Investigator — University of Oxford
Locations (1):
- John Radcliffe Hospital, Oxford, United Kingdom